CLINICAL TRIAL: NCT05214768
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Induction and Maintenance Study to Evaluate the Efficacy and Safety of CC-93538 in Adult and Adolescent Japanese Subjects With Eosinophilic Gastroenteritis
Brief Title: A Study to Evaluate the Efficacy and Safety of CC-93538 in Adult and Adolescent Japanese Participants With Eosinophilic Gastroenteritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-93538-EG-001
Record Dates: First submitted 2022-01-12; First posted 2022-01-31 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Eosinophilic Gastroenteritis
Keywords: Eosinophilic Gastroenteritis; CC-93538; Gastrointestinal Diseases; Eosinophilic Gastro-Intestinal Disorder; EGID; Digestive system diseases; Gastroenteritis
MeSH Terms: conditions — Eosinophilic enteropathy; Gastrointestinal Diseases; Digestive System Diseases; Gastroenteritis | interventions — cendakimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CC-93538 (Experimental)
  Interventions: Drug: CC-93538
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CC-93538 — Specified dose on specified days
  Other Names: Cendakimab; BMS-986355
  Arms: CC-93538
Drug: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of CC-93538 in adult and adolescent participants with eosinophilic gastroenteritis.

ELIGIBILITY:
Inclusion Criteria:

* Histologic evidence of eosinophilic gastroenteritis (EGE) defined as ≥ 30 eosinophils (eos)/high-power field (hpf) in at least 5 hpf in the stomach and/or ≥ 30 eos/hpf in at least 3 hpf in the duodenum while on stable background therapy for EGE
* Has weekly symptom scores of ≥ 4/15 for any of Gastric Pain Symptoms domain, Stomach Heaviness Symptom domains, and /or Diarrhea Symptoms domain as assessed by the Izumo Scale with electronic device for the 2 consecutive weeks before Day 1
* Must agree to maintain a stable diet from the first Screening Visit and throughout the duration of the study, and participants must have maintained a stable diet for at least 4 weeks prior to the first Screening Visit
* Females of childbearing potential must have 2 negative pregnancy tests as verified by the Investigator prior to starting study therapy and agree to practice a highly effective method of contraception until 5 months after the last dose

Exclusion Criteria:

* Ascites requiring treatment or symptomatic ascites
* History of inflammatory bowel disease, achalasia or esophageal surgery
* Has other causes of gastric and/or duodenal eosinophilia or eosinophilic granulomatosis with polyangiitis (EGPA)

Other protocol-defined inclusion/exclusion criteria apply

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2025-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (25):
- Japan (25):
  - Local Institution - 024, Gifu, Gifu
  - Local Institution - 022, Himeji-shi, Hyōgo
  - Local Institution - 009, Nishinomiya, Hyōgo
  - Local Institution - 0025, Tsu, Mie-ken
  - Local Institution - 025, Tsu, Mie-ken
  - Local Institution - 023, Sendai, Miyagi
  - Local Institution - 007, Bunkyo-ku, Tokyo
  - Local Institution - 001, Setagaya-ku, Tokyo
  - Local Institution - 010, Akita
  - Local Institution - 017, Hirosaki
  - Local Institution - 015, Hiroshima
  - Local Institution - 018, Kagoshima
  - Local Institution - 020, Kitakyushu
  - Local Institution - 004, Kobe
  - Local Institution - 011, Maebashi
  - Local Institution - 013, Nagaoka
  - Local Institution - 016, Nagasaki
  - Local Institution - 006, Nagoya
  - Local Institution - 021, Nagoya
  - Local Institution - 008, Niigata
  - Local Institution - 002, Osaka
  - Local Institution - 012, Ōgaki
  - Local Institution - 005, Shibukawa
  - Local Institution - 019, Tokyo
  - Local Institution - 003, Yamagata

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction Phase - CC-93538 360 mg QW: Participants with Eosinophilic Gastroenteritis received 360 mg CC-93538 subcutaneously (SC) once weekly in the induction phase.
- Induction Phase - Placebo: Participants with Eosinophilic Gastroenteritis received matching placebo once weekly in the induction phase.
- Maintenance Phase - CC-93538 360 mg QW: Participants with Eosinophilic Gastroenteritis received 360 mg CC-93538 subcutaneously (SC) once weekly in the maintenance phase.
- Maintenance Phase - CC-93538 360 QW/Q2W: Participants with Eosinophilic Gastroenteritis who were randomized to receive 360 mg CC-93538 once weekly in Induction Phase received CC-93538 360 mg SC once every other week for 32 weeks during Maintenance Phase.
- Maintenance Phase - Placebo: Participants with Eosinophilic Gastroenteritis received matching placebo once weekly in the maintenance phase.
- Open-Label Extension - CC-93538 360 mg QW: Participants with Eosinophilic Gastroenteritis received 360 mg CC-93538 subcutaneously (SC) once weekly in the open-label extension period.
Period: Induction Period
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo | Maintenance Phase - CC-93538 360 mg QW | Maintenance Phase - CC-93538 360 QW/Q2W | Maintenance Phase - Placebo | Open-Label Extension - CC-93538 360 mg QW
Started | 32 | 16 | 0 | 0 | 0 | 0
Completed | 30 (25 completed induction phase and 5 directly entered OLE phase) | 16 (12 completed induction phase and 4 directly entered OLE phase) | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Period
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo | Maintenance Phase - CC-93538 360 mg QW | Maintenance Phase - CC-93538 360 QW/Q2W | Maintenance Phase - Placebo | Open-Label Extension - CC-93538 360 mg QW
Started | 0 | 0 | 13 (2 out of 13 entered in OLE phase) | 12 (1 out of 12 entered in OLE phase) | 12 (1 out of 12 participant in OLE phase) | 0
Completed | 0 | 0 | 11 (All 11 participants entered OLE phase) | 10 (9 out of 10 participants entered OLE phase) | 11 (All 11 participants entered OLE phase) | 0
Not Completed | 0 | 0 | 2 | 2 | 1 | 0
Not completed — Other Reasons | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 1 | 0
Period: Open Label Extension Period
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo | Maintenance Phase - CC-93538 360 mg QW | Maintenance Phase - CC-93538 360 QW/Q2W | Maintenance Phase - Placebo | Open-Label Extension - CC-93538 360 mg QW
Started | 0 | 0 | 0 | 0 | 0 | 44 (9 participants from induction and 35 participants from maintenance entered in this arm.)
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 44
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Ongoing Study | 0 | 0 | 0 | 0 | 0 | 42

BASELINE CHARACTERISTICS:
Groups:
- CC-93538 360 mg QW: Participants with Eosinophilic Gastroenteritis received 360 mg CC-93538 subcutaneously (SC) once weekly in the induction phase and once weekly for 32 weeks in Maintenance Phase.
- Placebo: Participants with Eosinophilic Gastroenteritis received matching placebo once weekly in the induction phase and once weekly for 32 weeks in Maintenance Phase.
- Total: Total of all reporting groups
Arm/Group | CC-93538 360 mg QW | Placebo | Total
Number analyzed (Participants) | 32 | 16 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (16.79) | 41.8 (17.63) | 41.2 (16.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 18 | 10 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 32 | 16 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 32 | 16 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Number of Peak Eosinophils (Eos) Count Per High-power Field (Hpf) in Gastrointestinal (GI) Biopsies
Description: Blood samples were collected to assess eosinophils count. Baseline data are defined as last measurement collected on or prior the date of first dose for Induction Phase.
Time Frame: Baseline and Week 16
Population: Intent-to-treat (ITT) population which consists of all randomized participants regardless of whether or not the participant received IP (CC-93538 or placebo). Only participants analyzed at specified timepoint are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Peak # of eosinophils counted per field
Arm/Group | CC-93538 360 mg QW | Placebo
Number analyzed (Participants) | 30 | 16
Peak # of eosinophils counted per field | -100.4 (44.23) | 122.8 (60.27)
Statistical Analysis 1: Comparison: CC-93538 360 mg QW vs Placebo; Test type: Superiority; p = 0.003, ANCOVA; Least Square Mean Difference = -223.2, 95% CI 2-sided [-370.2 to -76.3], Standard Error of Mean 74.98

2. Secondary Outcome: Induction Phase: Changes in Each of 5 Domain Scores of the Izumo Scale From Baseline at Week 16
Description: The Izumo Scale questionnaire assesses the comprehensive 5 different GI symptom domains during the past week and consists with 15 weekly questions (3 questions per 1 domain): Heartburn Symptoms domain(Questions1 through3), Gastric Pain Symptoms domain(Questions4 through6), Stomach Heaviness Symptoms domain(Questions7 through9), Constipation Symptoms domain (Question 10 through12), Diarrhea Symptoms domain (Questions13 through15). Each question is scored on a 6-point Likert scale of "0 = No trouble at all" to "5 = Can't stand it," and the score for each question within a domain is added to determine domain specific scores scaled from 0 to 15, with higher values indicating greater symptom severity.
Time Frame: Baseline and Week 16
Population: Intent-to-treat (ITT) population which consists of all randomized participants regardless of whether or not the participant received IP (CC-93538 or placebo).
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | CC-93538 360 mg QW | Placebo
Number analyzed (Participants) | 32 | 16
Score on a Scale
  Heartburn Symptoms domain | -1.9 (0.46) | -1.7 (0.66)
  Gastric Pain Symptoms domain | -2.1 (0.60) | -0.9 (0.86)
  Stomach Heaviness Symptoms domain | -2.1 (0.61) | -2.2 (0.87)
  Constipation Symptoms domain | -1.0 (0.49) | -0.9 (0.69)
  Diarrhea Symptoms domain | -1.8 (0.46) | -1.6 (0.65)

3. Secondary Outcome: Induction + Maintenance: Changes in Each of 5 Domain Scores of the Izumo Scale From Baseline at Week 48
Description: The Izumo Scale questionnaire assesses the comprehensive 5 different GI symptom domains during the past week and consists with 15 weekly questions (3 questions per 1 domain): Heartburn Symptoms domain(Questions1 through3), Gastric Pain Symptoms domain(Questions4 through6), Stomach Heaviness Symptoms domain(Questions7 through9), Constipation Symptoms domain (Question 10 through12), Diarrhea Symptoms domain (Questions13 through15). Each question is scored on a 6-point Likert scale of "0 = No trouble at all" to "5 = Can't stand it," and the score for each question within a domain is added to determine domain specific scores scaled from 0 to 15, with higher values indicating greater symptom severity. Participants that discontinued Induction period without entering maintenance period are included in the CC-93538 360 mg QW arm.
Time Frame: Baseline and Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Groups:
- CC-93538 360 QW/Q2W: Participants with Eosinophilic Gastroenteritis who were randomized to receive 360 mg CC-93538 once weekly in Induction Phase received CC-93538 360 mg SC once every other week for 32 weeks during Maintenance Phase.
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W | Placebo
Number analyzed (Participants) | 20 | 12 | 16
Score on a Scale
  Heartburn Symptoms domain | 0.2 (0.74) | -2.0 (0.98) | -1.4 (0.84)
  Gastric Pain Symptoms domain | 0.1 (0.81) | -2.5 (1.08) | -1.8 (0.91)
  Stomach Heaviness Symptoms domain | 0.7 (0.81) | -3.4 (1.05) | -1.5 (0.90)
  Constipation Symptoms domain | 0.6 (0.79) | -1.0 (1.07) | -1.4 (0.85)
  Diarrhea Symptoms domain | 1.5 (0.87) | -0.1 (1.16) | -2.3 (0.97)

4. Secondary Outcome: Induction Phase: Percentage of Participants Who Achieve Both Clinical and Histologic Response Composite at Week 16
Description: Clinical response defined as percentage of participants who achieve <4/15 in each of three Symptoms of Interest (Gastric Pain Symptoms domain, Stomach Heaviness Symptoms domain, and Diarrhea Symptoms domain) scores of Izumo Scale from baseline. Histologic response defined as a > 75% reduction of peak gastric and/or duodenal eos count from baseline. Izumo Scale tests 5 different GI symptom domains during past week and consists with 15 weekly questions (3 questions per 1 domain): Heartburn Symptoms domain(Ques1 through3), Gastric Pain Symptoms domain(Questions4 through6), Stomach Heaviness Symptoms domain(Ques7 through9), Constipation Symptoms domain (Question 10 through12), Diarrhea Symptoms domain (Ques13 through15). Each question is scored on a 6-point Likert scale of "0 = No trouble at all" to "5 = Can't stand it," and score for each question within a domain added to determine domain specific scores scaled from 0 to 15, with higher values indicating greater symptom severity.
Time Frame: Week 16
Population: Intent-to-treat (ITT) population which consists of all randomized participants regardless of whether or not the subject received IP (CC-93538 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | CC-93538 360 mg QW | Placebo
Number analyzed (Participants) | 32 | 16
percentage of participants | 6.3 | 0

5. Secondary Outcome: Induction + Maintenance: Percentage of Participants Who Achieve Both Clinical and Histologic Response Composite at Week 48
Description: as for outcome 4
Time Frame: Baseline and week 48
Population: Intent-to-treat (ITT) population which consists of all randomized participants regardless of whether or not the subject received IP (CC-93538 or placebo). Only participants analyzed at specified timepoint are included in the analysis. Participants that discontinued Induction period without entering maintenance period are included in the CC-93538 360 mg QW arm.
Measure: Number; unit: percentage of participants
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W | Placebo
Number analyzed (Participants) | 20 | 12 | 16
percentage of participants | 0 | 8.3 | 0

6. Secondary Outcome: Induction + Maintenance: Change From Baseline in Mean Number of Peak Eosinophils (Eos) Count Per High-power Field (Hpf) in Gastrointestinal (GI) Biopsies at Week 48
Description: Blood samples were collected to assess eosinophils count. Baseline data are defined as last measurement collected on or prior the date of first dose for Induction Phase. Participants that discontinued Induction period without entering maintenance period are included in the CC-93538 360 mg QW arm
Time Frame: Baseline and Week 48
Population: Intent-to-treat (ITT) population which consists of all randomized participants regardless of whether or not the participant received IP (CC-93538 or placebo). Only participants with baseline measurements of peak eos analyzed at specified timepoint are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Peak # of eosinophils counted per field
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W | Placebo
Number analyzed (Participants) | 19 | 10 | 15
Peak # of eosinophils counted per field | -24.1 (61.26) | -151.2 (89.70) | 98.6 (66.03)

7. Secondary Outcome: Induction Phase: Percent Changes in Mean Number of Peak Eos Per Hpf in GI Biopsies From Baseline
Description: as for outcome 1
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | CC-93538 360 mg QW | Placebo
Number analyzed (Participants) | 30 | 16
Percent change | -13.4 (18.85) | 61.6 (22.18)

8. Secondary Outcome: Induction + Maintenance: Percent Changes in Mean Number of Peak Eos Per Hpf in GI Biopsies From Baseline
Description: as for outcome 6
Time Frame: Baseline and Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W | Placebo
Number analyzed (Participants) | 19 | 10 | 15
Percent change | 7.2 (29.78) | -39.9 (50.54) | 43.7 (36.15)

9. Secondary Outcome: Induction Phase: Percentage of Participants With Eosinophil Histologic Response (> 75% Reduction)
Description: Histologic response defined as a > 75% reduction of peak gastric and/or duodenal eos count from baseline.
Time Frame: Week 16
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | CC-93538 360 mg QW | Placebo
Number analyzed (Participants) | 32 | 16
percentage of participants | 15.6 | 0

10. Secondary Outcome: Induction + Maintenance: Percentage of Participants With Eosinophil Histologic Response (> 75% Reduction)
Description: Histologic response defined as a > 75% reduction of peak gastric and/or duodenal eos count from baseline. Participants that discontinued Induction period without entering maintenance period are included in the CC-93538 360 mg QW arm.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W | Placebo
Number analyzed (Participants) | 20 | 12 | 16
percentage of participants | 0 | 25.0 | 0

11. Secondary Outcome: Induction Phase: Percentage of Participants Who Achieve <4/15 in Each of Three Symptoms of Interest Scores Using the Izumo Scale
Description: The Izumo Scale questionnaire assesses the comprehensive 5 different GI symptom domains during the past week and consists with 15 weekly questions (3 questions per 1 domain): Heartburn Symptoms domain(Questions1 through3), Gastric Pain Symptoms domain(Questions4 through6), Stomach Heaviness Symptoms domain(Questions7 through9), Constipation Symptoms domain (Question 10 through12), Diarrhea Symptoms domain (Questions13 through15). Each question is scored on a 6-point Likert scale of "0 = No trouble at all" to "5 = Can't stand it," and the score for each question within a domain is added to determine domain specific scores scaled from 0 to 15, with higher values indicating greater symptom severity. Gastric Pain Symptoms domain, Stomach Heaviness Symptoms domain, and Diarrhea Symptoms domain are Symptoms of Interest.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | CC-93538 360 mg QW | Placebo
Number analyzed (Participants) | 32 | 16
percentage of participants | 28.1 | 18.8

12. Secondary Outcome: Induction + Maintenance: Percentage of Participants Who Achieve <4/15 in Each of Three Symptoms of Interest Scores Using the Izumo Scale
Description: The Izumo Scale questionnaire assesses the comprehensive 5 different GI symptom domains during the past week and consists with 15 weekly questions (3 questions per 1 domain): Heartburn Symptoms domain(Questions1 through3), Gastric Pain Symptoms domain(Questions4 through6), Stomach Heaviness Symptoms domain(Questions7 through9), Constipation Symptoms domain (Question 10 through12), Diarrhea Symptoms domain (Questions13 through15). Each question is scored on a scale of "0 = No trouble at all" to "5 = Can't stand it," and one symptom domain is scored from 0 to 15, with higher values indicating greater symptom severity. Gastric Pain Symptoms domain, Stomach Heaviness Symptoms domain, and Diarrhea Symptoms domain are Symptoms of Interest. Participants that discontinued Induction period without entering maintenance period are included in the CC-93538 360 mg QW arm. Only participants from ages 12 -19 years old at specified timepoint are included in the analysis.
Time Frame: Baseline and Week 48
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W | Placebo
Number analyzed (Participants) | 20 | 12 | 16
percentage of participants | 10.0 | 25.0 | 31.3

13. Secondary Outcome: Induction Phase: Changes in Total Score of Eosinophilic Gastrointestinal Disorder (EGID) Severity Score From Baseline to Weeks 16 in Adolescent (12 to 19 Years)
Description: The EGID Severity Score for participants from 12 to 19 years old assesses 6 different symptoms (vomiting, dysphagia, anorexia, abdominal pain, diarrhea, bloody stool), 2 clinical laboratory tests (albumin, eos ratio of peripheral blood cells) and general condition, including height and weight. The score ranges from 0 to 100 and the higher the score, the greater the severity. A score of ≥ 40 is considered as severe, a score of 15 to 39 as moderate and ≤ 14 score as mild.
Time Frame: Baseline and Week 16
Population: Intent-to-treat (ITT) population which consists of all randomized participants regardless of whether or not the subject received IP (CC-93538 or placebo). Only participants analyzed at specified timepoint are included in the analysis. Only participants from ages 12 -19 years old at specified timepoint are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | CC-93538 360 mg QW | Placebo
Number analyzed (Participants) | 5 | 3
Score on a Scale | -6.4 (1.70) | -3.8 (2.91)

14. Secondary Outcome: Induction Phase: Changes in Total Score of EGID Severity Score From Baseline to Weeks 16 in Adults (>= 20 Years)
Description: The EGID Severity Scores are assessed by the investigator. The EGID Severity Score for participants ≥ 20 years old assess the intensity and the frequency of 6 different symptoms (vomiting, dysphagia, anorexia, abdominal pain, diarrhea, bloody stool), 2 clinical laboratory tests (albumin, eos ratio of peripheral blood cells) and 2 medical history items (history of surgery and use of systemic corticosteroid or immunosuppressives). The score ranges from 0 to 82 and the higher the score, the greater the severity. A score of ≥ 40 is considered as severe, a score of 15 to 39 as moderate and a score of ≤ 14 score as mild.
Time Frame: Baseline and Week 16
Population: Intent-to-treat (ITT) population which consists of all randomized participants regardless of whether or not the subject received IP (CC-93538 or placebo). Only participants analyzed at specified at specified timepoint are included in the analysis. Only participants from ages >=20 years years old at specified timepoint are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | CC-93538 360 mg QW | Placebo
Number analyzed (Participants) | 25 | 11
Score on a Scale | -5.5 (1.40) | -4.5 (2.12)

15. Secondary Outcome: Induction+ Maintenance: Changes in Total Score of EGID Severity Score From Baseline to Weeks 48 in Adolescent (12 to 19 Years)
Description: The EGID Severity Score for participants from 12 to 19 years old assesses 6 different symptoms (vomiting, dysphagia, anorexia, abdominal pain, diarrhea, bloody stool), 2 clinical laboratory tests (albumin, eos ratio of peripheral blood cells) and general condition, including height and weight. The score ranges from 0 to 100 and the higher the score, the greater the severity. A score of ≥ 40 is considered as severe, a score of 15 to 39 as moderate and ≤ 14 score as mild. Participants that discontinued Induction period without entering maintenance period are included in the CC-93538 360 mg QW arm.
Time Frame: Baseline and Week 48
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W | Placebo
Number analyzed (Participants) | 2 | 2 | 1
Score on a Scale | 7.1 (0.00) | -10.4 (0.00) | 1.7 (0.00)

16. Secondary Outcome: Induction + Maintenance: Changes in Total Score of EGID Severity Score From Baseline to Weeks 48 in Adults (>= 20 Years)
Description: The EGID Severity Scores are assessed by the investigator. The EGID Severity Score for participants ≥ 20 years old assess the intensity and the frequency of 6 different symptoms (vomiting, dysphagia, anorexia, abdominal pain, diarrhea, bloody stool), 2 clinical laboratory tests (albumin, eos ratio of peripheral blood cells) and 2 medical history items (history of surgery and use of systemic corticosteroid or immunosuppressives). The score ranges from 0 to 82 and the higher the score, the greater the severity. A score of ≥ 40 is considered as severe, a score of 15 to 39 as moderate and a score of ≤ 14 score as mild. Participants that discontinued Induction period without entering maintenance period are included in the CC-93538 360 mg QW arm.
Time Frame: Baseline and Week 48
Population: Intent-to-treat (ITT) population which consists of all randomized participants regardless of whether or not the subject received IP (CC-93538 or placebo). Only participants analyzed at specified timepoint are included in the analysis. Only participants from ages >=20 years old at specified timepoint are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W | Placebo
Number analyzed (Participants) | 14 | 4 | 9
Score on a Scale | -3.3 (2.76) | -2.4 (5.32) | -7.2 (3.35)

17. Secondary Outcome: Induction Phase: Time to First Event of Eosinophilic Gastroenteritis (EGE) Flare and First Use of Rescue Therapy
Description: Any worsening of EGE symptoms during study participation will be documented as an EGE flare. Worsening of EGE symptoms is defined as continuous worsening of symptoms for 2 consecutive visits (4 weeks apart) compared to baseline, measured by the weekly Izumo Scale score (≥ 4 weeks of no change from baseline or ≥ 4 weeks of worsening from baseline).
Time Frame: Through Week 16
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CC-93538 360 mg QW | Placebo
Number analyzed (Participants) | 32 | 16
days
  EGE Flare | NA [NA to NA] — Not estimated due to insufficient number of events | NA [113 to NA] — Not estimated due to insufficient number of events
  Use of rescue therapy | NA [NA to NA] — Not estimated due to insufficient number of events | NA [113 to NA] — Not estimated due to insufficient number of events

18. Secondary Outcome: Induction + Maintenance: Time to First Event of Eosinophilic Gastroenteritis (EGE) Flare and First Use of Rescue Therapy
Description: Any worsening of EGE symptoms during study participation will be documented as an EGE flare. Worsening of EGE symptoms is defined as continuous worsening of symptoms for 2 consecutive visits (4 weeks apart) compared to baseline, measured by the weekly Izumo Scale score (≥ 4 weeks of no change from baseline or ≥ 4 weeks of worsening from baseline). Participants that discontinued Induction period without entering maintenance period are included in the CC-93538 360 mg QW arm.
Time Frame: Through Week 48
Population: Intent-to-treat (ITT) population which consists of all randomized participants regardless of whether or not the subject received IP (CC-93538 or placebo). Only participants analyzed at specified timepoint are included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W | Placebo
Number analyzed (Participants) | 20 | 12 | 16
days
  EGE Flare | NA [92 to NA] — Not estimated due to insufficient number of events | NA [NA to NA] — Not estimated due to insufficient number of events | NA [113 to NA] — Not estimated due to insufficient number of events
  Use of rescue therapy | NA [113 to NA] — Not estimated due to insufficient number of events | NA [NA to NA] — Not estimated due to insufficient number of events | NA [115 to NA] — Not estimated due to insufficient number of events

19. Secondary Outcome: Maintenance Phase: Time to Reduce to Zero Concomitant Corticosteroid Use
Description: Participants who use concomitant corticosteroid at baseline and entered Maintenance Phase
Time Frame: From Week 16 through Week 48
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W | Placebo
Number analyzed (Participants) | 7 | 4 | 6
days | NA [144 to NA] — Not estimated due to insufficient number of events | NA [176 to NA] — Not estimated due to insufficient number of events | NA [113 to NA] — Not estimated due to insufficient number of events

20. Secondary Outcome: Percentage of Participants for Whom the Dose of Concomitant Steroids is Reduced to Zero
Description: Participants who use concomitant corticosteroid at baseline and entered Maintenance period were included in the analysis.
Time Frame: Week 24, 32, 40 and 48
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W | Placebo
Number analyzed (Participants) | 7 | 4 | 6
percentage of participants
  Week 24 | 0 | 0 | 0
  Week 32 | 0 | 0 | 0
  Week 40 | 14.3 | 0 | 0
  Week 48 | 14.3 | 25.0 | 0

21. Secondary Outcome: Induction and Maintenance: Number of Participants With Treatment-Emergent Adverse Events
Description: A treatment emergent adverse event (TEAE) is any AE that emerges during treatment or Safety Follow-up Period having been absent pre-treatment or worsens in severity relative to the pretreatment state. Participants that discontinued Induction period without entering maintenance period are included in the CC-93538 360 mg QW arm.
Time Frame: From Day 1 untill Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W | Placebo
Number analyzed (Participants) | 20 | 12 | 16
Participants
  Any TEAEs | 16 | 9 | 13
  Any Serious TEAEs | 0 | 1 | 0
  Any Moderate or Severe TEAE | 10 | 6 | 10
  ANY TEAE suspected to be related to study drug | 6 | 3 | 2

22. Secondary Outcome: Induction and Maintenance: Number of Participants With Remarkable Differences of Clinically Relevant Mean Changes From Baseline in Vital Signs Measurements
Description: Participants that discontinued Induction period without entering maintenance period are included in the CC-93538 360 mg QW arm.
Time Frame: From Day 1 untill Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W | Placebo
Number analyzed (Participants) | 20 | 12 | 16
Participants | 0 | 0 | 0

23. Secondary Outcome: Induction and Maintenance: Number of Participants With Remarkable Differences of Clinically Relevant Mean Changes From Baseline in Physical Examinations Parameters
Description: as for outcome 22
Time Frame: From Day 1 untill Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W | Placebo
Number analyzed (Participants) | 20 | 12 | 16
Participants | 0 | 0 | 0

24. Secondary Outcome: Induction and Maintenance: Number of Participants With Mean Changes Over Time That Were of Clinically Concern in Hematology Parameters, Serum Chemistry Parameters, and Urinalysis Parameters
Description: as for outcome 22
Time Frame: From Day 1 untill Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W | Placebo
Number analyzed (Participants) | 20 | 12 | 16
Participants | 0 | 0 | 0

25. Secondary Outcome: Induction and Maintenance: Number of Participants With Anti-Drug-Antibody
Description: Blood samples were collected to assess Anti-Drug-Antibody. Participants that discontinued Induction period without entering maintenance period are included in the CC-93538 360 mg QW arm.
Time Frame: From Day 1 till Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W
Number analyzed (Participants) | 20 | 12
Participants | 2 | 0

26. Secondary Outcome: Induction Phase: CC-93538 Trough Concentration at Week 16
Description: Blood samples were collected to assess CC-93538 trough concentrations.
Time Frame: Week 16
Population: Pharmacokinetic population included all participants who received at least one dose of active drug and have at least one measurable concentration data. Only participants with data available at specified timepoint and receiving CC-93538 were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | CC-93538 360 mg QW
Number analyzed (Participants) | 30
ng/mL | 179472.2 (47.2)

27. Secondary Outcome: Maintenance Phase: CC-93538 Trough Concentration at Week 48
Description: Blood samples were collected to assess CC-93538 trough concentrations. Participants that discontinued Induction period without entering maintenance period are included in the CC-93538 360 mg QW arm.
Time Frame: Week 48
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | CC-93538 360 mg QW | CC-93538 360 QW/Q2W
Number analyzed (Participants) | 9 | 7
ng/mL | 165591.7 (58.5) | 76433.4 (64.1)

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious and non-serious adverse events were collected from first dose (day 1) and up to 121 weeks.
Description: All-cause mortality, serious and non-serious adverse events were collected for all participants who received at least one dose of IP. As pre-specified adverse events for participants that discontinued Induction period without entering maintenance period were collected in the CC-93538 360 mg QW arm.
Groups:
- Induction and Maintenance - CC-93538 360mg QW: Participants with Eosinophilic Gastroenteritis received 360 mg CC-93538 subcutaneously (SC) once weekly in the induction phase and once weekly for 32 weeks in Maintenance Phase.
- Maintenance - CC-93538 360mg QW/Q2W: Participants with Eosinophilic Gastroenteritis who were randomized to receive 360 mg CC-93538 once weekly in Induction Phase received CC-93538 360 mg SC once every other week for 32 weeks during Maintenance Phase.
- Induction and Maintenance - Placebo: Participants with Eosinophilic Gastroenteritis received matching placebo once weekly in the induction phase and once weekly for 32 weeks in Maintenance Phase.
- Open-label Long-term Extension Phase - CC-93538 360mg QW: Participants with Eosinophilic Gastroenteritis earlier randomized to Induction and Maintenance phase received 360 mg CC-93538 subcutaneously (SC) once weekly in Open-Label Long-term Extension phase.
Arm/Group | Induction and Maintenance - CC-93538 360mg QW | Maintenance - CC-93538 360mg QW/Q2W | Induction and Maintenance - Placebo | Open-label Long-term Extension Phase - CC-93538 360mg QW
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/12 | 0/16 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/12 | 0/16 | 0/44
Other Adverse Events (participants affected / at risk) | 16/20 | 9/12 | 13/16 | 30/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction and Maintenance - CC-93538 360mg QW (N=20) | Maintenance - CC-93538 360mg QW/Q2W (N=12) | Induction and Maintenance - Placebo (N=16) | Open-label Long-term Extension Phase - CC-93538 360mg QW (N=44)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction and Maintenance - CC-93538 360mg QW (N=20) | Maintenance - CC-93538 360mg QW/Q2W (N=12) | Induction and Maintenance - Placebo (N=16) | Open-label Long-term Extension Phase - CC-93538 360mg QW (N=44)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Cataract (Eye disorders) | 1 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 2
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Iritis (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 2
Fatigue (General disorders) | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 5 | 2 | 1 | 5
Malaise (General disorders) | 0 | 0 | 1 | 2
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 4 | 3
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1 | 0 | 0
Food allergy (Immune system disorders) | 1 | 0 | 0 | 1
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 2
COVID-19 (Infections and infestations) | 2 | 4 | 0 | 8
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 1 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1 | 6
Nasopharyngitis (Infections and infestations) | 1 | 6 | 3 | 4
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 1
Perineal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 2
Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Eosinophil count increased (Investigations) | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Essential tremor (Nervous system disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 3
Migraine (Nervous system disorders) | 0 | 0 | 2 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Eosinophilic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
NSAID exacerbated respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT05214768/Prot_SAP_000.pdf